CLINICAL TRIAL: NCT06398158
Title: Clinical and Radiological Outcomes in People With Aquaporin-4 IgG Positive Neuromyelitis Optica Spectrum Disorder Treated With Ravulizumab
Brief Title: Study of the Clinical and Radiological Impact of Ravulizumab in People With Neuromyelitis Optica Spectrum Disorder
Acronym: AMAZE
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Darin Okuda, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2023-0744
Record Dates: First submitted 2024-04-16; First posted 2024-05-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Neuromyelitis Optica
MeSH Terms: conditions — Neuromyelitis Optica | interventions — ravulizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be routinely collected during the course of the study, in addition to acute clinical relapses to assess the temporal course of change in serum neurofilament light chain, glial fibrillary acidic protein, tau, and ubiquitin carboxyl-terminal hydrolase levels.
  Data captured from the samples collected may be utilized in the future to identify or verify putative prognostic and predictive markers associated with disease and markers of therapeutic response to treatment. Baseline and dynamic (within study) clinical disease characteristics and associated biomarker data may be utilized to predict subsequent disease advancement along with severity, identifying high-risk subgroups and identify predictors of response to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- NMOSD: 35 people with aquaporin-4 IgG antibody positive neuromyelitis optica spectrum disorder is planned with all individuals treated with commercially supplied ravulizumab at the recommendation of the healthcare provider, with use consistent with the approved indication and labeling. Approximately 50% of the cohort is anticipated to be Black/African American based on existing internal data.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — All study participants will receive commercially covered ravulizumab consistent with the indication, dose and frequency contained within the approved label.

SUMMARY:
This is an observational study to:

* evaluate the on-treatment clinical performance of ravulizumab in relation to the pre-treatment time period (time period prior to exposure),
* enhance knowledge regarding conventional MRI outcomes in people with NMOSD treated with ravulizumab,
* identify factors suggestive of subclinical disease progression through conventional MRI sequences,
* determine if treatment with ravulizumab, impacts longitudinal 3D conformational MRI measures at the dorsal medulla and other regions of the CNS, and
* identify biomarkers (e.g., serum neurofilament light chain (sNfL), conventional and novel MRI markers, etc.) related to disease activity.

DETAILED DESCRIPTION:
This is a single-center prospective observational study with all participants recruited from The University of Texas Southwestern Medical Center in Dallas, Texas. Enrollment of 35 people with aquaporin-4 IgG antibody positive neuromyelitis optica spectrum disorder is planned with all individuals treated with commercially supplied ravulizumab at the recommendation of the healthcare provider, with use consistent with the approved indication and labeling.

The study is composed of the following:

1. Study screening: Study screening will occur up to 45 days, with a minimum of 3 days to allow for the scheduling of study related events. During this time the eligibility of participants will be evaluated and diagnosis of aquaporin 4-IgG positive neuromyelitis optica spectrum confirmed by both the Core Clinical Committee and Core Imaging Committee. If a subject is declared a screen failure, all reasons for ineligibility will be captured. Ineligible subjects may be rescreened at a later time.
2. Open-label treatment with commercially covered ravulizumab: Enrolled subjects will be treated with ravulizumab in a manner consistent with the FDA approved labeling. All prescreening laboratory tests, vaccinations, and clinical surveillance studies will be ordered and managed by the Primary Clinical Team.

   Treatment with ravulizumab will continue throughout the course of the study unless one of the following events occur: a. An individual loses commercial coverage for ravulizumab; b. Discontinuation of the medication by the clinical team is recommended due to an adverse reaction, intolerability, or inadequate disease control. The decision regarding treatment will be determined by the Primary Clinical Team and the patient; c. The participant prematurely discontinues treatment for personal reasons

   In the event that the medication is discontinued prematurely, participants will continue to be followed throughout the 52-78 week period with all clinical, radiological, and serological assessments performed.
3. Clinical surveillance: Clinical safety surveillance will be performed throughout the study and managed by the Primary Clinical Team. In the event of new or concerning clinical symptoms, participants will be evaluated within a 24-hour period via telehealth or in-person visit. Clinical evaluations, serological assessments, and repeat MRI data per protocol will be performed within a 48-hour period. The acute management of subjects will be led by the Primary Clinical Team. All clinical data associated with acute clinical events will be sent to the Core Clinical Committee and relapses adjudicated by consensus. MRI data acquired at the time of the event will be evaluated by the Core Imaging Committee and interval change in conventional imaging outcomes (i.e., new and/or newly enlarging T2-hyperintense lesions, gadolinium enhancement) adjudicated by consensus.
4. Safety surveillance: Safety assessments in association with treatment with ravulizumab will be managed by the Primary Clinical Team. The use of concomitant medications will be tracked during the entire course of the study. These will include prescribed medications for both NMOSD and non-NMOSD, including the use of glucocorticosteroid treatment administered orally or parenterally, along with over-the-counter agents.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent available prior to conduct of any study associated activities
2. Men and women > 18 years of age
3. Aquaporin-4 IgG positive people with neuromyelitis optica spectrum disorder treated with commercially available ravulizumab in a manner consistent with the approved indication
4. Expanded Disability Status Scale score of <7.0

Exclusion Criteria:

1. Individuals who are intolerant to MRI
2. Individuals previously exposed to eculizumab with treatment discontinuation due to lack of effective disease control (i.e., clinical relapse or demonstration of MRI advancement after 12 weeks of sustained treatment exposure)
3. Unresolved meningococcal disease
4. History of an active infection
5. Existing participation in neuromyelitis optical spectrum disorder interventional clinical studies
6. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female adult participants recruited from The Multiple Sclerosis and Neuroimmunology Clinic at The University of Texas Southwestern Medical Center in Dallas, Texas.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical relapses before and after treatment with ravulizumab | 52 weeks - 78 weeks
  Compare the number of participants with adjudicated clinical relapses both pre- and post-ravulizumab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Darin T. Okuda, MD, Principal Investigator — University of Texas Southwestern Medical Center; Peter Sguigna, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No